CLINICAL TRIAL: NCT01418560
Title: Renal Sympathetic Modification in Patients With Chronic Renal Failure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Second Affiliated Hospital of Chongqing Medical University (Other)
Collaborators: Jiangsu Provincial People's Hospital (Other); Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Yuehui Yin, Director and Professor, Dept. of Cardiology, the second affiliated hospital of Chongqing Medical University, Chongqing Cardiac arrhythmias service center, The Second Affiliated Hospital of Chongqing Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SWAN-RF
Record Dates: First submitted 2011-08-15; First posted 2011-08-17 (Estimated); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Chronic Renal Failure
Keywords: renal artery; sympathetic nerves; modification; chronic renal failure
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- renal sympathetic modification (Experimental): Renal artery ablation to modify sympathetic activity in patients with chronic renal failure.
  Interventions: Procedure: renal sympathetic modification
- Absolute medicine therapy (No Intervention): Maintenance of anti-renal failure medications only

INTERVENTIONS:
Procedure: renal sympathetic modification — Device: THERMOCOOL® Catheter Renal sympathetic modification with a catheter-based procedure
  Other Names: renal denervation
  Arms: renal sympathetic modification

SUMMARY:
The purpose of this study is to observe the incident of uremia and dialysis requirement after renal sympathetic modification using THERMOCOOL® catheter in patients with chronic renal failure, and evaluate safety and efficacy of the intervention.

DETAILED DESCRIPTION:
Chronic renal failure is serial clinical manifestations because of kidney damage. Previous studies found sympathetic nerves over activity in chronic renal failure patients. Traditional therapies included medications and dialysis replacement therapy need to spend much money. Renal ablation for sympathetic modification is a new method which is proved to be effective in decreasing sympathetic nerves activity. We assume that modifying renal sympathetic activity by ablation is effective and safe in treatment of chronic renal failure. This trial is going to recruit 200 patients (Ablation group VS Control group = 1:1) with a follow-up duration of 3 years. Patients in ablation group will receive additional necessary medications besides expectant intervention, and patients in control group will receive appropriate medications only. We aim to observe the effect of serum creatinine, creatinine clearance rate, glomerular filtration rate, urine microalbumin, urine microalbumin/creatinine, and composite cardio cerebrovascular events after renal sympathetic modification using THERMOCOOL® catheter, and evaluate safety and efficacy of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old, and ≤ 75 years old of age
* at least three months history of definite kidney damage
* renal function of serum creatinine of < 354umol/L, and/or creatinine clearance rate of ≥ 30ml/min, and/or estimated glomerular filtration rate of ≥ 45ml/min for recent 2-3 times evaluation. Besides, the value of creatinine clearance rate fluctuated no more than 30% in recent three months, and 15% in the following two weeks.
* urine microalbumin, and/or urine microalbumin/creatinine is abnormal, and/or quantity of 24 hrs urine protein suggests kidney damage.
* is competent and willing to provide written, informed consent to participate in this clinical study

Exclusion Criteria:

* congenital renal diseases cause to chronic renal damage
* estimated glomerular filtration rate (eGFR) of < 45mL/min
* taking medicine of glucocorticosteroids, non-steroid anti-inflammatory drugs (NSAIDs), or cytotoxic drugs at present
* value of 24 hrs urine protein is of > 10g at least once in recent three months, or serum albumin of < 25g/L
* has the history of renal restenosis or renal stents implantation
* has experienced AMI (old myocardial infarction is not excluded), unstable angina pectoris, cerebrovascular accidents, and alimentary tract hemorrhage within 3 months
* carcinoma patients
* patients with sick sinus syndrome
* pregnant women
* mental disorders
* patients that have allergy to contrast agent
* patients that do not go with follow-up
* others such as researcher considers it is not appropriate to be included into the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2011-08 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
the incident of uremia and dialysis requirement | three years

SECONDARY OUTCOMES:
serum creatinine increases into multiples in 1 month follow-up | three years
effect of urine microalbumin, urine microalbumin/creatinine, serum creatinine, or 24 hrs urine protein value | three years
incidence of composite cardiovascular events | three years

CONTACTS AND LOCATIONS:
Locations (1):
- 2ndChongqingMU, Chongqing, Chongqing Municipality, China